CLINICAL TRIAL: NCT05331859
Title: Topical Insulin Versus Autologous Serum and Enhanced Corneal Epithelial Healing After Keratorefractive Surgeries
Brief Title: Topical Insulin Versus Autologous Serum After Corneal Surgeries
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Taher Eleiwa, Dr, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TIKRS
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Corneal Epithelial Wound
Keywords: lasik; PRK; topical insulin; autologous serum
MeSH Terms: interventions — Insulin; Congresses as Topic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional (Placebo Comparator): Corneal epithelial wound healing in patients who received photorefractive keratectomy (PRK) treated only with conventional postoperative eye drops.
  Interventions: Drug: conventional
- Insulin (Active Comparator): Corneal epithelial wound healing in patients who received photorefractive keratectomy (PRK) treated with topical insulin and conventional postoperative eye drops.
  Interventions: Drug: Insulin; Drug: conventional
- Autologous serum eye drops (Active Comparator): Corneal epithelial wound healing in patients who received photorefractive keratectomy (PRK) treated with Autologous serum eye and conventional postoperative eye drops.
  Interventions: Drug: autologous serum (AS); Drug: conventional

INTERVENTIONS:
Drug: Insulin — Topical insulin drops will be prepared by diluting 1 unit of rapid-acting insulin per 1 mL of an artificial tear with a propylene glycol base. Drops will be preserved at low temperature (2ºC) and applied four times a day.
  Arms: Insulin
Drug: autologous serum (AS) — Whole blood (20 ml) wll be procured by venipuncture, centrifuged at 1,500 revolutions per minute (relative centrifugal force of 25.15 × g) for 10 minutes. AS drops will be carefully prepared under a laminar airflow cabinet, and diluted with artificial tears (Systane ultra; Alcon) to 20%. AS drops will be prepared on the day of surgery and patients will be asked to keep AS drops refrigerated at about 4C.
  Arms: Autologous serum eye drops
Drug: conventional — Topical moxifloxacin 0.5% (Vigamox; Alcon Laboratories) four times per day, artificial tears (Systane ultra; Alcon) every two hours, Dexamethasone 0.1% (Maxidex; Alcon Laboratories) four times daily for one month then fluorometholone 0.1% (Efemyo; Orchidia Laboratories) four times daily for another two to four weeks depending on refraction and haze level.

SUMMARY:
The aim of the study is to test whether use of topical insulin or autologous serum eye-drops can promote corneal epithelial healing following photorefractive keratectomy (PRK).

DETAILED DESCRIPTION:
Topical insulin has been proved recently to enhance the corneal reepithelization rate and manage neurotrophic corneal ulcers unresponsive to conventional treatments. However, its effectiveness on corneal epithelial wound healing in patients who received photorefractive keratectomy (PRK) has not been reported. In this study, we plan to perform a prospective non-randomized study to determine the efficacy and safety of topical insulin as a primary treatment for a corneal epithelial defect in patients undergoing the PRK and compare that to autologous serum eye drops. The study eye will receive either the insulin or the serum eye drops, in addition to the conventional treatment, while the control eye will have the standard treatment. For each eligible candidate, the eye with a higher depth of ablation will be the study eye. If even ablation depth in both eyes, the right eye will be selected. The conventional postoperative eye drops include topical moxifloxacin 0.5% (Vigamox; Alcon Laboratories) four times per day, artificial tears (Systane Ultra; Alcon) every two hours, Dexamethasone 0.1% (Maxidex; Alcon Laboratories) four times daily for one month followed by fluorometholone 0.1% (Efemyo; OrchidiaLaboratories) four times daily for another two to four weeks depending on refraction and haze level. In study eyes, the patients receive either topical insulin eye drops or autologous serum in addition to conventional postoperative eye drops until complete epithelial healing. The duration for the corneal surface to completely re-epithelize, the grade of postoperative corneal haze, the incidence of corneal complications due to delayed surface re-epithelization (e.g. infectious corneal ulcer, corneal melting, sterile corneal ulcer, corneal neovascularization), and the distant corrected visual acuity will be compared between these three groups.

ELIGIBILITY:
Inclusion Criteria:

* stable refraction of at least one year, normal corneal topography, and a minimum central corneal thickness of 500 μm.

Exclusion Criteria:

* unstable refraction, dry eye, blepharitis, corneal disease, glaucoma, systemic diseases including infectious and collagen vascular diseases, diabetes, and topographical evidence of keratoconus.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Duration for the corneal surface to completely re-epithelialize. | up to 6 weeks
Grade of postoperative corneal haze | 6 weeks
  0, completely clear cornea; +0.5, barely visible corneal opacity; +1, reticular subepithelial opacities not interfering with visibility of fine iris details; +2, punctate or coalesced subepithelial opacities with mild obscuration of iris details; +3, confluent subepithelial opacities with moderate obscuration of the iris and lens; and +4, dense opacities with complete opacification of the stroma.

SECONDARY OUTCOMES:
Incidence of corneal complications due to delayed surface re-epithelization (e.g. infectious corneal ulcer, sterile corneal ulcer, corneal melting, corneal neovascularization). | 6 weeks
Best-corrected Visual Acuity improvement (Snellen, decimal) | Before and after treatment completion, assessed up to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Taher Eleiwa, MD PhD, Principal Investigator — Benha University
Locations (2):
- Egypt (2):
  - Ebsar Eye Centre, Banhā, Kalyobeya
  - Benha University, Banhā

IPD SHARING:
Plan to Share IPD: Yes
The completed data will be shared upon a reasonable request to the principal investigator.
Supporting Information: Study Protocol, CSR
Time Frame: For 1 year after the publishing the results

REFERENCES:
- [Result] Diaz-Valle D, Burgos-Blasco B, Rego-Lorca D, Puebla-Garcia V, Perez-Garcia P, Benitez-Del-Castillo JM, Herrero-Vanrell R, Vicario-de-la-Torre M, Gegundez-Fernandez JA. Comparison of the efficacy of topical insulin with autologous serum eye drops in persistent epithelial defects of the cornea. Acta Ophthalmol. 2022 Jun;100(4):e912-e919. doi: 10.1111/aos.14997. Epub 2021 Aug 18. PMID 34407296
- [Result] Diaz-Valle D, Burgos-Blasco B, Gegundez-Fernandez JA, Garcia-Caride S, Puebla-Garcia V, Pena-Urbina P, Benitez-Del-Castillo JM. Topical insulin for refractory persistent corneal epithelial defects. Eur J Ophthalmol. 2021 Sep;31(5):2280-2286. doi: 10.1177/1120672120958307. Epub 2020 Sep 21. PMID 32951459
- [Result] Akcam HT, Unlu M, Karaca EE, Yazici H, Aydin B, Hondur AM. Autologous serum eye-drops and enhanced epithelial healing time after photorefractive keratectomy. Clin Exp Optom. 2018 Jan;101(1):34-37. doi: 10.1111/cxo.12574. Epub 2017 Jul 18. PMID 28718904